CLINICAL TRIAL: NCT04385576
Title: Taiwan "Aerosol Box" Versus UMMC "Intubation Box" : Clinical Evaluation of the "Intubation Box" for Ease of Intubation
Brief Title: Taiwan "Aerosol Box" Versus UMMC "Intubation Box"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr SHAIRIL RAHAYU BINTI RUSLAN, Clinical Lecturer, University of Malaya
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2020410-8498
Record Dates: First submitted 2020-04-28; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Airway
Keywords: intubation box; COVID-19; personnel protective equipment
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerosol Box (Active Comparator): Intubation using the Taiwan model Aerosol Box to assess the duration of time needed for successful endotracheal intubation of an airway manikin.
  Interventions: Device: Aerosol Box; Device: Intubation Box
- Intubation Box (Active Comparator): Intubation using the UMMC model Intubation Box to assess the duration of time needed for successful endotracheal intubation of an airway manikin.
  Interventions: Device: Aerosol Box; Device: Intubation Box

INTERVENTIONS:
Device: Aerosol Box — Usage of an Intubation Box to minimize intubator and environment contamination during intubation and extubation. Time taken for first-pass success if also expected to be reduced with the usage of the Intubation Box.
Device: Intubation Box — Usage of an Intubation Box to minimize intubator and environment contamination during intubation and extubation. Time taken for first-pass success if also expected to be reduced with the usage of the Intubation Box.

SUMMARY:
This study compares two intubation boxes, that is the Taiwan "Aerosol Box" versus the UMMC "Intubation Box". The importance of this intubation box has come to light recently in view of the COVID-19 pandemic and the fact that intubation is an aerosol-generating procedure. Risks of the healthcare worker attending to the airway of COVID-19 patients is high and the intubation box aims to minimize that and reduce contamination of the environment. The original design of the "Aerosol Box" has limitations and is not easily used by intubators. This study evaluates the clinical usefulness of an innovation of the "Aerosol Box" design that is made to be more ergonomic and increases the rate of successful intubation. Anaesthetists with more than 5 years of clinical experience in intubating airways as well as more than 20 successful intubations using videolaryngoscopy , will be available to participate. This study will employ manikin and will be a randomized cross-over trial, conducted in UM.

DETAILED DESCRIPTION:
Background:

Intubation is classified as an aerosol-generating procedure (AGP). Intubation in a confirmed COVID-19 patient with a high viral load poses a high risk of exposure to health care workers (HCW). To reduce this risk, the HCW and their assistants are advised to don full personnel protective equipment (PPE) with a powered air purifying respiratory (PAPR) during intubation. In view of this concern, this procedure is highly recommended to be done in a negative pressure room to control the spread of aerosolizing particles in the room. A first-pass success in intubation is also crucial to minimize the risk of infection to health care workers involved.

Introduction :

An Aerosol Box (from here on known as Box A) was recently designed by Dr. Lai Hsien Yung from Taiwan which adds extra protection to the intubator and the surrounding environment. The Aerosol Box is a transparent box made of acrylic or transparent polycarbonate sheet, designed with an opening on one side allowing it to fit over the patient's chest and neck, while the opposing side has two holes through which the intubator can insert their hands through. It was shown that this barrier enclosure during intubation protects the laryngoscopist. A recent study simulated a patient with a cough during intubation with and without the Aerosol Box. With the box, it was demonstrated that the simulated cough resulted in contamination of only the inner surface of the box, the laryngoscopist's gloves and gowned forearms. Examination of the laryngoscopist and the room with ultraviolet light after the simulated cough also showed no macroscopic contamination outside the box. In contrast, intubation without the box demonstrated that the laryngoscopist's gown, gloves, face mask, eye shield, hair, neck, ears, and shoes were all contaminated.

Feedbacks from our colleagues stated that intubation with Box A is slightly difficult and may cause delay in intubation. Canelli et al also concluded this observation. The investigators, therefore, innovated the design of Box A to facilitate the laryngoscopist, known as the UMMC Intubation Box (from here on known as Box B).

ELIGIBILITY:
Inclusion Criteria:

* anaesthetists with more than 5 years of clinical experience AND more than 20 successful intubations using a videolaryngoscope

Exclusion Criteria:

* anaesthetists with less than 5 years of clinical experience AND/OR less than 20 successful intubations using a videolaryngoscope

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2020-09-15 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to successful intubation | 10 minutes
  The interval from insertion of the laryngoscope blade into the mouth to inflation of the tracheal tube cuff

SECONDARY OUTCOMES:
Number of intubation attempts | 10 minutes
  Number of attempts taken to successfully intubate the airway manikin
Evaluation of the intubator's experience using both boxes | 10 minutes
  Evaluation of the intubator's experience using both boxes using a questionnaire based on the ISO9421-11 standard, that is effectiveness, efficiency and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: INA I SHARIFFUDDIN, MAnaes, Study Director — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Selangor, Malaysia

REFERENCES:
- [Result] Canelli R, Connor CW, Gonzalez M, Nozari A, Ortega R. Barrier Enclosure during Endotracheal Intubation. N Engl J Med. 2020 May 14;382(20):1957-1958. doi: 10.1056/NEJMc2007589. Epub 2020 Apr 3. No abstract available. PMID 32243118
- See also: Taiwanese doctor invents device to protect US doctors against coronavirus — https://www.taiwannews.com.tw/en/news/3902435

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT04385576/Prot_SAP_ICF_000.pdf